CLINICAL TRIAL: NCT02560220
Title: A Single-arm Phase-I Trial for the Determination of Safety and Feasibility of the Intravenous Administration of Mitomycin C-treated Donor Peripheral Blood Mononuclear Cells (MICs) for Individualized Immunosuppression in Living Donor Kidney Transplant Recipients (TOL-1 Study)
Brief Title: MIC Cell Therapy for Individualized Immunosuppression in Living Donor Kidney Transplant Recipients
Acronym: TOL-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: WiSP GmbH (Other); German Federal Ministry of Economics and Technology (Other Government)
Responsible Party: Principal Investigator, Christian Morath, M.D., Martin Zeier, M. D., Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TOL-1
Record Dates: First submitted 2015-08-06; First posted 2015-09-25 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention arm (Experimental): Patients receive MIC cell therapy together with standard immunosuppressive therapy
  Interventions: Biological: Mitomycin C-induced peripheral blood mononuclear cells (MICs)

INTERVENTIONS:
Biological: Mitomycin C-induced peripheral blood mononuclear cells (MICs) — MICs are given intravenously 2 or 7 days before kidney transplantation from a living donor

SUMMARY:
A phase- I clinical trial to determine safety and feasibilty of intravenous administration of mitomycin C-treated donor peripheral blood mononuclear cells in patients with chronic kidney disease stage KDIGO 4 or 5 (i.e. GFR 15-30 mL/min or < 15 mL/min) who receive a kidney transplant from a living donor.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage KDIGO 4 or 5
* First kidney transplant from a living donor
* Age ≥ 18 years
* ABO compatible
* CDC-PRA < 20%
* No donor-specific antibodies
* Negative CDC and ELISA crossmatch
* Immunosuppression with cyclosporin A, EC-MPS and methylprednisolone
* Informed consent
* Adequate contraception (women with child bearing potential)

Exclusion Criteria:

* Psychiatric disorder
* Heart failure (NYHA III or IV)
* Severe liver disease
* Active hepatitis B or C or HIV infection
* Active bacterial, fungal or viral disease
* Malignancy or malignancy in the last 5 years before screening
* Preexisting immunosuppression
* Vaccination with a live vaccine in the last 3 months before screening
* S/p splenectomy
* Substance abuse
* Pregnancy or lactation
* Women: Child/pregnancy with the intended donor
* Allergy against the investigational drug or part of it
* Other diseases that prohibit participation in the study (in the opinion of the investigator)
* Participation in an other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the frequency of adverse events after intravenous administration of MICs within 30 days after transplantation. | 30 days

SECONDARY OUTCOMES:
Cumulative incidence of infection | 30 days
Cumulative incidence of CMV reactivation | 30 days
Number of patients with PTLD | 30 days
Number of patients with delayed graft function | 7 days
Number of patients with a pos. CDC and/or ELISA crossmatch | day -1 before transplantation
Number of patients with DSA | day -1 before transplantation and day 7 and 30 after transplantation
Incidence of biopsy-proven cellular rejection | 30 days
Incidence of biopsy-proven antibody-mediated rejection | 30 days
Number of patients with stable graft function (S-creatinine < 2mg/dL) | 30 days
Patient and graft survival | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zeier, MD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Morath C, Schmitt A, Zeier M, Schmitt M, Sandra-Petrescu F, Opelz G, Terness P, Schaier M, Kleist C. Cell therapy for immunosuppression after kidney transplantation. Langenbecks Arch Surg. 2015 Jul;400(5):541-50. doi: 10.1007/s00423-015-1313-z. Epub 2015 Jun 17. PMID 26077202
- [Background] Kleist C, Sandra-Petrescu F, Jiga L, Dittmar L, Mohr E, Greil J, Mier W, Becker LE, Lang P, Opelz G, Terness P. Generation of suppressive blood cells for control of allograft rejection. Clin Sci (Lond). 2015 May;128(9):593-607. doi: 10.1042/CS20140258. PMID 25495457
- [Background] Dittmar L, Mohr E, Kleist C, Ehser S, Demirdizen H, Sandra-Petrescu F, Hundemer M, Opelz G, Terness P. Immunosuppressive properties of mitomycin C-incubated human myeloid blood cells (MIC) in vitro. Hum Immunol. 2015 Jul;76(7):480-7. doi: 10.1016/j.humimm.2015.06.008. Epub 2015 Jun 11. PMID 26074415
- [Background] Terness P, Oelert T, Ehser S, Chuang JJ, Lahdou I, Kleist C, Velten F, Hammerling GJ, Arnold B, Opelz G. Mitomycin C-treated dendritic cells inactivate autoreactive T cells: toward the development of a tolerogenic vaccine in autoimmune diseases. Proc Natl Acad Sci U S A. 2008 Nov 25;105(47):18442-7. doi: 10.1073/pnas.0807185105. Epub 2008 Nov 18. PMID 19017789
- [Derived] Schaier M, Morath C, Wang L, Kleist C, Opelz G, Tran TH, Scherer S, Pham L, Ekpoom N, Susal C, Ponath G, Kalble F, Speer C, Benning L, Nusshag C, Mahler CF, Pego da Silva L, Sommerer C, Huckelhoven-Krauss A, Czock D, Mehrabi A, Schwab C, Waldherr R, Schnitzler P, Merle U, Schwenger V, Krautter M, Kemmner S, Fischereder M, Stangl M, Hauser IA, Kalsch AI, Kramer BK, Bohmig GA, Muller-Tidow C, Reiser J, Zeier M, Schmitt M, Terness P, Schmitt A, Daniel V. Five-year follow-up of a phase I trial of donor-derived modified immune cell infusion in kidney transplantation. Front Immunol. 2023 Jul 11;14:1089664. doi: 10.3389/fimmu.2023.1089664. eCollection 2023. PMID 37483623
- [Derived] Morath C, Schaier M, Ibrahim E, Wang L, Kleist C, Opelz G, Susal C, Ponath G, Aly M, Alvarez CM, Kalble F, Speer C, Benning L, Nusshag C, Pego da Silva L, Sommerer C, Huckelhoven-Krauss A, Czock D, Mehrabi A, Schwab C, Waldherr R, Schnitzler P, Merle U, Tran TH, Scherer S, Bohmig GA, Muller-Tidow C, Reiser J, Zeier M, Schmitt M, Terness P, Schmitt A, Daniel V. Induction of Long-Lasting Regulatory B Lymphocytes by Modified Immune Cells in Kidney Transplant Recipients. J Am Soc Nephrol. 2023 Jan 1;34(1):160-174. doi: 10.1681/ASN.2022020210. Epub 2022 Sep 22. PMID 36137752
- [Derived] Morath C, Schmitt A, Kleist C, Daniel V, Opelz G, Susal C, Ibrahim E, Kalble F, Speer C, Nusshag C, Pego da Silva L, Sommerer C, Wang L, Ni M, Huckelhoven-Krauss A, Czock D, Merle U, Mehrabi A, Sander A, Hackbusch M, Eckert C, Waldherr R, Schnitzler P, Muller-Tidow C, Hoheisel JD, Mustafa SA, Alhamdani MS, Bauer AS, Reiser J, Zeier M, Schmitt M, Schaier M, Terness P. Phase I trial of donor-derived modified immune cell infusion in kidney transplantation. J Clin Invest. 2020 May 1;130(5):2364-2376. doi: 10.1172/JCI133595. PMID 31990685